CLINICAL TRIAL: NCT06503874
Title: Intensive Attention Training to Treat Brain Fog in Individuals With Long-Covid
Brief Title: Improving Attention in Individuals With Long COVID-19
Acronym: LongCovAtten
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Shira Cohen-Zimerman, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00220499; 90IFDV0033-01-00 (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Long Covid
Keywords: COVID-19; Brain Fog
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Mental Fatigue

STUDY DESIGN:
Intervention Model Description: First, participants will complete the pre-treatment assessment. Participants then will be randomized to either immediate APT-3 group, delayed APT or Music activity group.
  The interventions (APT-3 or Music activity) will last 4 weeks. At the end of the intervention participants will undergo another assessment battery, and once again at 1-month post intervention follow-up.
  Following the maintenance assessment, participants from the Music activity group will have the option to receive the APT-3 intervention. If they accept, they will undergo another assessment battery at the end of the 4-week intervention.
  Participants from the delayed APT-3 group will undergo the week 5 assessment and will then be offered to enroll in the APT-3 training. If they accept, they will undergo another assessment battery at the end of the 4-week intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Training (Experimental): The computer based APT-3 intervention will be delivered in a hybrid model that will combine in-person therapy sessions at Shirley Ryan AbilityLab and practice sessions which will be completed remotely. The dosing of each intervention training will be 30 minutes per day, 5 days a week, for 4 weeks (10 hours total over 4 weeks). The difficulty of the tasks in both interventions will increase progressively as the participants improve in their skills. APT-3 treatment will be administered by a trained and certified speech-language pathologist.
  Interventions: Other: Attention Training
- Music Program (Experimental): This group will receive an enhanced music experience. They will listen to pre determined music for 30 minutes per day, 5 days a week, for 4 weeks (10 hours total over 4 weeks). This will be delivered in a hybrid model that will combine, in person, remote, and independent sessions, similar to the Attention Training group. Once they complete the music program, they will have the option to complete the Attention Training.
  Interventions: Other: Music Group
- Delayed Attention Training (No Intervention): This group will not be provided any program for the initial 4 weeks. After they complete the week 5 assessments, they will have the option to complete the Attention Training.

INTERVENTIONS:
Other: Attention Training — The APT-3 is an evidence-based, standardized computer-based training program that was designed to improve attention skills that underlie higher level cognitive processes (e.g., executive functions and memory).
  Other Names: APT-3
  Arms: Attention Training
Other: Music Group — This group will listen to a pre-determined playlist of music following the same dosing as the attention training group as stated in the arms.
  Arms: Music Program

SUMMARY:
This study is to find out if the Attention Processing Training program is a potential treatment for brain fog symptoms, reported by people with Long-Covid. Also investigating the feasibility of completing this program virtually.

DETAILED DESCRIPTION:
The goal of this project is to test the feasibility, acceptability and efficacy of an attention training intervention (Attention Process Training; APT-3) as a potential treatment for brain fog symptoms experienced by people with Long-Covid. There already is good empirical evidence to support the idea that the APT-3 treatment is feasible and effective in improving attention in people with acquired brain injuries, but information about its efficacy and acceptability in people with Long-Covid brain fog is lacking.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years. Live in the Chicagoland area
* A history of confirmed SARS-CoV-2 infection.
* Subjective reports of cognitive symptoms that interfere with everyday activities, starting on or shortly after SARS-CoV-2 infection.
* Continuation or development of Long-Covid brain fog 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation.
* Objective attentional deficits as measured by the Conners CPT-312, and/or the Digit Span subtest (WAIS- III13).
* Able to use a keyboard.
* Able to understand and communicate in English.
* Able to consent independently.

Exclusion Criteria:

* Being hospitalized due to COVID-19 diagnosis for more than 3 days.
* Pre-morbid neurological conditions that could potentially affect cognition, such as Parkinson's Disease, Alzheimer's Dementia, acquired brain injury.
* Severe depression.
* Currently enrolled in cognitive training or physical exercise training.
* Receiving chemotherapy or radiation within last 6 months.
* Active substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who successfully completed at least 80% of the study tasks sessions | 2 years
  Recording the number of participants who completed at least 80% of the study sessions out of the number of all participants who enrolled in the study.

SECONDARY OUTCOMES:
Change of scores in objective attention tests (i.e, CPT 3), pre- and post -intervention | 2 year
  The Conners Continuous Performance Test Third Edition™ (Conners CPT 3™)

OTHER OUTCOMES:
Change of scores in objective attention tests (i.e, Digit Span), pre- and post -intervention | 2 year
  Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) - Digit Span Subtest

CONTACTS AND LOCATIONS:
Overall Officials: Shira Cohen-Zimerman, PhD, Principal Investigator — Shirley Ryan AbilityLab; Elliot Roth, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States